CLINICAL TRIAL: NCT04963439
Title: A Single-center, Open-label, Single-dose, Randomized, 2-way Crossover Phase 1 Study in Healthy Adult Participants to Assess the Relative Oral Bioavailability of Two Macitentan Pediatric Formulations
Brief Title: A Study of Two Macitentan Pediatric Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR109027; 2021-001258-67 (EudraCT Number); 67896062PAH1008 (Other: Actelion)
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive single oral dose of macitentan formulated as final market image (FMI) in fasted conditions (test) (Treatment A) in treatment period 1 followed by a single oral dose of macitentan as the clinical service formulation (CSF) in fasted conditions (reference) (Treatment B) in treatment period 2 on Day 1. Study intervention intake in subsequent intervention periods in an individual participant will be separated by a washout period of at least 10 days.
  Interventions: Drug: Macitentan
- Treatment Sequence BA (Experimental): Participants will receive Treatment B in treatment period 1 followed by Treatment A in treatment period 2 on Day 1. Study intervention intake in subsequent intervention periods in an individual participant will be separated by a washout period of at least 10 days.
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan dispersible tablets will be administered orally as per assigned treatment sequence.
  Other Names: Opsumit; ACT-064992

SUMMARY:
The purpose of this study is to assess the rate and extent of absorption of macitentan following administration of a single oral dose of macitentan formulated as final market image (FMI) (test), compared to macitentan as the clinical service formulation (CSF) under fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical and surgical history collected at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Systolic blood pressure (SBP) between 100 and 145 millimeters of mercury (mmHg) (inclusive) and diastolic blood pressure (DBP) between 50 and 90 mmHg (inclusive) at screening, preferably measured on the right arm, supine after 5 minutes of rest and standing after 3 minutes
* Twelve-lead electrocardiogram (ECG) with heart rate between 45 and 90 beats per minute (bpm) and without clinically relevant abnormalities, at the discretion of the investigator, measured after the participant is supine for at least 5 minutes, at screening
* Body weight not less than 50.0 kilograms (kg) and body mass index (BMI) between 18.5 and 30.0 kilograms per meter square (kg/m^2) (inclusive)
* All women must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta- hCG]) pregnancy test at screening and must have a negative urine pregnancy test on Day -1 of each intervention period

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to macitentan or drugs of the same class, or any excipients of the drug formulations
* Taken any disallowed therapies, concomitant therapy within 14 days (or longer, based on elimination half-life) before administration of study intervention in the first intervention period
* Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 30 days or 10 half-lives (whichever is longer) before study intervention intake in the first intervention period, or received a biological product within 3 months or 10 half-lives (whichever is longer) before study intervention intake in the first intervention period, or is currently enrolled in an investigational study
* Values of hepatic aminotransferase (alanine aminotransferase and/or aspartate aminotransferase) greater than (>) 1.5 * upper limit of normal at screening
* Positive results from the human immunodeficiency virus (HIV) (type 1 and 2) serology at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Macitentan | Predose and up to 216 hours post dose (Up to Day 10)
  Cmax is defined as maximum observed plasma analyte concentration of Macitentan.
Area Under the Plasma Analyte Concentration-time Curve of Macitentan from Time Zero to Time of the Last Quantifiable Concentration (AUC [0-last]) | Predose and up to 216 hours post dose (Up to Day 10)
  AUC (0-last) is defined as area under the plasma analyte concentration-time curve of macitentan from time zero to time of the last quantifiable (non-below quantification limit [BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Analyte Concentration-time Curve of Macitentan from Time Zero to Infinity (AUC [0-infinity]) | Predose and up to 216 hours post dose (Up to Day 10)
  AUC (0-infinity) is defined as area under the plasma analyte concentration-time curve of macitentan from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), where AUC (0-last) is area under the plasma analyte concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) plasma analyte concentration and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Actual Sampling Time to Reach the Maximum Observed Plasma Analyte Concentration (Tmax) of Macitentan and its Metabolite ACT-132577 | Predose and up to 216 hours post dose (Up to Day 10)
  Tmax is defined as actual sampling time to reach the maximum observed plasma analyte concentration of macitentan and its metabolite ACT-132577.
Last Observed Measurable Plasma Analyte Concentration (Clast) of Macitentan and its Metabolite ACT-132577 | Predose and up to 216 hours post dose (Up to Day 10)
  Clast is defined as last observed measurable BQL plasma analyte concentration of macitentan and its metabolite ACT-132577.
Area Under the Plasma Analyte Concentration-time Curve of Macitentan and its Metabolite ACT-132577 from Time Zero to 72 Hours (AUC [0-72 Hours]) Postdose | Predose up to 72 hours post dose
  AUC (0-72 hours) is defined as area under the plasma analyte concentration-time curve of macitentan and its metabolite ACT-132577 from time zero to 72 hours postdose, calculated by linear-linear trapezoidal summation.
Apparent Terminal Elimination Half-life (t1/2) of Macitentan and its Metabolite ACT-132577 | Predose and up to 216 hours post dose (Up to Day 10)
  t1/2 of macitentan and its metabolite ACT-132577 is time measured for the plasma analyte concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Apparent Terminal Elimination Rate Constant (Lambda[z]) of Macitentan and its Metabolite ACT-132577 | Predose and up to 216 hours post dose (Up to Day 10)
  Lambda(z) of macitentan and its metabolite ACT-132577 is defined as apparent terminal elimination rate constant, estimated by linear regression using the terminal log-linear phase of the log transformed concentration versus time curve.
Total Apparent Oral Clearance (CL/F) of Macitentan and its Metabolite ACT-132577 | Predose and up to 216 hours post dose (Up to Day 10)
  CL/F of macitentan and its metabolite ACT-132577 is defined as total apparent oral clearance, calculated as dose/AUC (0-infinity).
Apparent Volume of Distribution (Vdz/F) of Macitentan and its Metabolite | Predose and up to 216 hours post dose (Up to Day 10)
  Vdz/F of macitentan and its metabolite ACT-132577 is defined as apparent volume of distribution, calculated as dose/(Lambda[z]*AUC [0-infinity]).
Maximum Observed Plasma Analyte Concentration (Cmax) of Metabolite ACT-132577 | Predose and up to 216 hours post dose (Up to Day 10)
  Cmax is defined as maximum observed plasma analyte concentration of metabolite ACT-132577.
Area Under the Plasma Analyte Concentration-Time Curve of Metabolite ACT-132577 from Time Zero to Time of the Last Quantifiable Concentration (AUC [0-last]) | Predose and up to 216 hours post dose (Up to Day 10)
  AUC (0-last) of metabolite ACT-132577 is defined as area under the plasma analyte concentration-time curve from time zero to time of the last quantifiable (BQL) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Analyte Concentration-Time Curve of Metabolite ACT-132577 from Time Zero to Infinity (AUC [0-infinity]) | Predose and up to 216 hours post dose (Up to Day 10)
  AUC (0-infinity) is defined as area under the plasma analyte concentration-time curve of metabolite ACT-132577 from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), where AUC (0-last) is area under the plasma analyte concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) plasma analyte concentration and lambda(z) is apparent terminal elimination rate constant.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 10
  AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. SAE is any untoward medical occurrence that at any dose may results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Number of Participants with Abnormalities in Physical Examination | Up to Day 10 of each treatment period (Up to 7 weeks)
  Number of participants with abnormalities in physical examination (including general appearance, respiratory, neurological, eyes, ear/nose/throat, thyroid, cardiovascular, abdominal/gastrointestinal, hepatic, musculoskeletal, and dermatologic) will be reported.
Number of Participants with Abnormalities in Vital Signs | Up to Day 10 of each treatment period (Up to 7 weeks)
  Number of participants with abnormalities in vital signs (including temperature [tympanic], pulse rate, and blood pressure) will be reported.
Number of Participants with Abnormalities in Electrocardiograms (ECGs) | Up to Day 10 of each treatment period (Up to 7 weeks)
  Number of participants with abnormalities in ECGs will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to Day 10 of each treatment period (Up to 7 weeks)
  Number of participants with abnormalities in clinical laboratory tests (such as serum chemistry, hematology, and urinalysis) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency